CLINICAL TRIAL: NCT05705076
Title: Efficacy of Direct Oral Anticoagulants as a Prophylactic Anticoagulation of Catheter Induced Thrombosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R.22.10.1907.R1.R2.R3
Record Dates: First submitted 2023-01-21; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Anticoagulants; Increased

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo without anticoagulation (Placebo Comparator): Without any anticoagulation
  Interventions: Drug: catheter induced thromboprophylaxis
- Low Dose Direct Oral Anticoagulation (Active Comparator): Apixaban 2.5 mg twice Rivaroxaban 10 mg plus placebo
  Interventions: Drug: catheter induced thromboprophylaxis

INTERVENTIONS:
Drug: catheter induced thromboprophylaxis — Direct oral anticoagulation for catheter induced thromboprophylaxis

SUMMARY:
Direct Oral Anticoagulants

INTRODUCTION:

DOAC's looks like an attractive alternative to VKA because they offer important advantages beyond their easiness of administration, like less interactions and no need of laboratory monitoring. 1 All oral anticoagulant regimens but not aspirin were associated with a lower risk of recurrent VTE, while only VKAs were associated with a higher risk of major bleeding. 2 There have been significant differences between VKAs and DOACs in the risk of major bleeding by the current study size. Even though the risk of major bleeding with VKAs may be lower in patients already challenged to anticoagulation treatment. 3 Furthermore, when deciding on longer term secondary prevention of VTE, DOACs appeared safer than standard-intensity VKAs, taking clinically relevant bleeding or any bleeding into consideration.4-5 Until now there is no randomized controlled trial assessing the role of oral direct anticoagulant as a prophylaxis for catheter associated venous thromboembolism.

Aim of the work: To evaluate the efficacy of direct oral anticoagulants as a prophylactic anticoagulation in thromboprophylaxis of catheter induced thrombosis.

Patients and methods Study location: The study will be conducted at the department of vascular surgery in Mansoura University, Faculty of Medicine, Mansoura, Egypt .

Type of study: Randomized Controlled Prospective study Study duration: 2 years: 2022-2024 Sample size: It will include all patients presented to our department fulfilling the inclusion criteria.

Study population: The study will be conducted in patients with any permanent catheter inserted intravenous either femoral or jugular either for hemodialysis or replacement therapy .

Inclusion criteria: Any permanent catheter inserted intravenous either femoral or jugular either for hemodialysis, replacement or chemotherapy.

Exclusion criteria: History of central venous occlusion, contraindication of direct oral anticoagulants.

Consent: Patients must sign informed consent about possible complications from the therapy.

Data collection: The demographics, symptoms, and preoperative clinical data will be collected.

History Data: including underlying medical conditions, any previous associated morbidity.

Examination: Venous examinations. Laboratory: Blood picture, Blood sugar level, Kidney functions, Liver functions and Coagulation profile.

Imaging: Duplex US Method of Randomization: Computer-based Therapies group A : Apixaban 2.5 mg twice group B : Rivaroxaban 10 mg plus placebo group C : Placebo without anticoagulation Follow up All patients are followed by duplex ultrasonography to assess the thrombosis at the tip of catheter or around the catheter 10 days postoperative and 1, 3, 6, months then after one year, venography is indicated if the clinical evaluation not matched with sonographic results.

DETAILED DESCRIPTION:
INTRODUCTION:

DOAC's looks like an attractive alternative to VKA because they offer important advantages beyond their easiness of administration, like less interactions and no need of laboratory monitoring. 1 All oral anticoagulant regimens but not aspirin were associated with a lower risk of recurrent VTE, while only VKAs were associated with a higher risk of major bleeding. 2 There have been significant differences between VKAs and DOACs in the risk of major bleeding by the current study size. Even though the risk of major bleeding with VKAs may be lower in patients already challenged to anticoagulation treatment. 3 Furthermore, when deciding on longer term secondary prevention of VTE, DOACs appeared safer than standard-intensity VKAs, taking clinically relevant bleeding or any bleeding into consideration.4-5 Until now there is no randomized controlled trial assessing the role of oral direct anticoagulant as a prophylaxis for catheter associated venous thromboembolism.

Aim of the work: To evaluate the efficacy of direct oral anticoagulants as a prophylactic anticoagulation in thromboprophylaxis of catheter induced thrombosis.

Patients and methods Study location: The study will be conducted at the department of vascular surgery in Mansoura University, Faculty of Medicine, Mansoura, Egypt .

Type of study: Randomized Controlled Prospective study Study duration: 2 years: 2022-2024 Sample size: It will include all patients presented to our department fulfilling the inclusion criteria.

Study population: The study will be conducted in patients with any permanent catheter inserted intravenous either femoral or jugular either for hemodialysis or replacement therapy .

Inclusion criteria: Any permanent catheter inserted intravenous either femoral or jugular either for hemodialysis, replacement or chemotherapy.

Exclusion criteria: History of central venous occlusion, contraindication of direct oral anticoagulants.

Consent: Patients must sign informed consent about possible complications from the therapy.

Data collection: The demographics, symptoms, and preoperative clinical data will be collected.

History Data: including underlying medical conditions, any previous associated morbidity.

Examination: Venous examinations. Laboratory: Blood picture, Blood sugar level, Kidney functions, Liver functions and Coagulation profile.

Imaging: Duplex US Method of Randomization: Computer-based Therapies Group A : Apixaban 2.5 mg twice Group B : Rivaroxaban 10 mg plus placebo Group C : Placebo without anticoagulation Follow up All patients are followed by duplex ultrasonography to assess the thrombosis at the tip of catheter or around the catheter 10 days postoperative and 1, 3, 6, months then after one year, venography is indicated if the clinical evaluation not matched with sonographic results.

Statistical analysis

· The data will be analyzed using Statistical Package for the Social Sciences. The numerical outcomes e.g. age is calculated as mean. Gender will be recorded as frequency and percentage. Chi Square test is applied to assess the association of various parameters. The results will be considered statistically significant if the p-value is found to be less than or equal to 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Any permanent catheter inserted intravenous either femoral or jugular either for hemodialysis, replacement or chemotherapy.

Exclusion Criteria:

* History of central venous occlusion, contraindication of direct oral anticoagulants.

Ages: 10 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2023-01-24 (Estimated); Primary Completion 2024-03-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
thromboprophylaxis of catheter induced thrombosis | 6 months
  Prevention of thrombosis

SECONDARY OUTCOMES:
Duplex ultrasonography | 6 months
  duplex ultrasonography of central venous system

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593